CLINICAL TRIAL: NCT05278780
Title: Medication Abortion With Autonomous Self-Assessment Project: Pilot Study
Brief Title: Medication Abortion With Autonomous Self-Assessment Project
Acronym: MA-ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Stanford University (Other); Planned Parenthood of the Rocky Mountains (Unknown); Planned Parenthood North Central States (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1054
Record Dates: First submitted 2022-02-24; First posted 2022-03-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2023-03

CONDITIONS: Abortion Early
MeSH Terms: interventions — Mass Screening; Eligibility Determination

STUDY DESIGN:
Intervention Model Description: Case series study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Asynchronous screening (Experimental): Participants will be screened for medication abortion eligibility using written or online materials and questionnaires, without a synchronous conversation between the prescribing clinician and the patient.
  Interventions: Other: Screening for eligibility

INTERVENTIONS:
Other: Screening for eligibility — Asynchronous screening

SUMMARY:
In this study, the investigators propose to create and pilot-test an asynchronous medication abortion provision service.

DETAILED DESCRIPTION:
In this study, the investigators propose to create and pilot-test an asynchronous medication abortion (MA) provision service. The foundation of this service will be a website that provides information combined with a linked screening questionnaire. The questionnaire will be designed to collect the information recommended by current MA guidelines for history-based MA eligibility assessment. If the patient's responses meet specified criteria, the questionnaire will be sent to a study clinician, who will then determine whether a real-time clinical consultation or facility-based tests are needed. If the clinician decides that they are not, treatment will be provided accordingly. The primary goal of the study is to collect preliminary data on feasibility of the approach, abortion outcomes, and participant satisfaction. The investigators will use these data to determine whether to proceed with further development of asynchronous MA provision.

ELIGIBILITY:
Inclusion Criteria:

* • Has reviewed the study website

  * Can speak and read English
  * Has an address in a state where the study clinicians are licensed to practice medicine and where the service is legal
  * Is at least 18 years old
  * Is pregnant with a gestational age of ≤54 days from last menstrual period
  * Desires MA
  * Has not had an ultrasound in the current pregnancy (see below)
  * Has no symptoms of or risk factors for ectopic pregnancy
  * Has no medical contraindications to MA, specifically:

    * Hemorrhagic disorder or concurrent anticoagulant therapy
    * Chronic adrenal failure
    * Concurrent long-term systemic corticosteroid therapy
    * Inherited porphyria
    * Allergy to mifepristone or misoprostol, or other prostaglandin
  * Is comfortable obtaining the abortion pills without a pre-treatment ultrasound and without speaking by phone or video with the abortion provider.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  Proportion of treated participants with SAE (serious adverse effects) related to the study

SECONDARY OUTCOMES:
Incidence of participant questions | 12 months
  The proportion of participants who have questions after completing the questionnaire

OTHER OUTCOMES:
Proportion of participants who liked the service | 12 months
  Participant satisfaction upon exiting study evaluated using a participant satisfaction survey questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Planned Parenthood of the Rocky Mountains, Boulder, Colorado
  - Planned Parenthood North Central States, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No